CLINICAL TRIAL: NCT05487586
Title: Real-World Study of Ceftazidime-Avibactam to Characterize the Usage in Clinical Practice
Brief Title: Real-World Study of Ceftazidime Avibactam in China
Acronym: REACT
Status: Terminated | Type: Observational
Why Stopped: The study was prematurely discontinued due to slow enrollment and strategic considerations. This decision was not based on any safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3591037
Record Dates: First submitted 2022-07-11; First posted 2022-08-04 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hospital Acquired Pneumonia; Ventilator Acquired Pneumonia; Complicated Intra Abdominal Infections
Keywords: hospital acquired pneumonia; ventilator acquired pneumonia; complicated intra abdominal infections; ceftazidime avibactam; carbapenem-resistant Enterobacteriaceae
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ceftazidime avibactam group: Receive ≥1 dose of ceftazidime avibactam in routine practice; Aged ≥ 18 years old at the time of the informed consent signature.
  Interventions: Drug: ceftazidime avibactam group

INTERVENTIONS:
Drug: ceftazidime avibactam group — Non-Interventional Study
  Other Names: CAZ/AVI group

SUMMARY:
This observational study will enroll approximately 450 in patients. Patients treated with CAZ AVI for at least 1 dose at around 20 research centers in China will be enroll.

DETAILED DESCRIPTION:
The recruitment will last for approximately 6 months or until recruitment target is met, and information about treatment will be collected from the patients' medical records. Patients will be followed from CAZ AVI initiation until death, withdraw of the study, 60 days after discharged from the hospitalization, whichever comes first. The endpoint events will be evaluated at: 7 days, 14 days, 21 days, 30 days, 60 days, and end of treatment (EOT) after CAZ AVI initiation, if patients are not discharged prior to the next upcoming timepoint; and 30 days, 60 days after discharge.

ELIGIBILITY:
Inclusion criteria：

* Initiate ≥1 dose of ceftazidime-avibactam during hospitalization.
* Aged ≥ 18 years old at the time of the informed consent signature.
* Provide signed informed consent. Exclusion criteria：
* Are enrolled in any clinical trial, including enrollment in non interventional studies.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients treated with CAZ AVI for ≥1 dose in approximately 20 study sites.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- China (17):
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The First affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - The Affiliated People's Hospital of Ningbo University, Ningbo
  - Shanghai Tenth People's Hospital, Shanghai
  - The Second People's Hospital of Hebei Medical University, Shijiazhuang
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjing
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who received at least one dose of ceftazidime-avibactam during hospitalization were enrolled. Participants were recruited across 15 clinical research centers in China and were followed from first dose of ceftazidime-avibactam until death, withdrawal from study or 60 days post hospital discharge, whichever occurred first. Participants who initiated treatment with >=1 dose of ceftazidime-avibactam from 01 July 2022 to 31 December 2022 (index period of 6 months) were enrolled.
Pre-assignment Details: Data was abstracted from medical records and evaluated over approximately 21 months of this study.
Groups:
- Ceftazidime-Avibactam: Eligible participants who received at least one dose of ceftazidime-avibactam during hospitalization were enrolled in this study.
Period: Overall Study
Arm/Group | Ceftazidime-Avibactam
Started | 220
Completed | 192
Not Completed | 28
Not completed — Death | 22
Not completed — Physician Decision | 1
Not completed — Transfer to another hospital | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (16.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 150
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success Rate at Day 7
Description: The clinical success rate was defined as the number of participants with clinical outcome as "success" in a specific visit / number of participants with clinical outcome assessed in a specific visit and was reported in terms of percentage of participants. Clinical outcome as success was defined as resolution of all signs and symptoms of infection such that no further antimicrobial therapy was necessary. 95% CI was based on Clopper-Pearson method.
Time Frame: Day 7 (from the data evaluated in approximately 21 months of the study)
Population: The clinically evaluable (CE) analysis set included all participants from the full analysis set (FAS) with at least 72 hours use of ceftazidime-avibactam and at least 1 non-missing clinical evaluation outcome. The FAS included all enrolled participants. The enrolled participants met the inclusion criteria, and did not meet the exclusion criteria. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 153
Percentage of Participants | 37.3 [29.6 to 45.4]

2. Primary Outcome: Clinical Success Rate at Day 14
Description: as for outcome 1
Time Frame: Day 14 (from the data evaluated in approximately 21 months of the study)
Population: The CE analysis set included all participants from the FAS with at least 72 hours use of ceftazidime-avibactam and at least 1 non-missing clinical evaluation outcome. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 125
Percentage of Participants | 44.8 [35.9 to 54.0]

3. Primary Outcome: Clinical Success Rate at Day 21
Description: as for outcome 1
Time Frame: Day 21 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 94
Percentage of Participants | 46.8 [36.4 to 57.4]

4. Primary Outcome: Clinical Success Rate at Day 30
Description: as for outcome 1
Time Frame: Day 30 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 69
Percentage of Participants | 43.5 [31.6 to 56.0]

5. Primary Outcome: Clinical Success Rate at Day 60
Description: as for outcome 1
Time Frame: Day 60 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 29
Percentage of Participants | 69.0 [49.2 to 84.7]

6. Primary Outcome: Clinical Success Rate at End of Treatment (EOT)
Description: as for outcome 1
Time Frame: At EOT (maximum 86 days of treatment exposure) (from the data evaluated in approximately 21 months of the study)
Population: The CE analysis set included all participants from the FAS with at least 72 hours use of ceftazidime-avibactam and at least 1 non-missing clinical evaluation outcome.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Percentage of Participants | 66.4 [59.6 to 72.7]

7. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Site Investigator at Day 7
Description: The microbiological success rate was defined as the number of participants with microbiological outcome "success" in a specific visit / number of participants with microbiological outcome assessed in a specific visit and was reported in terms of percentage of participants. Microbiological outcome as success was defined as absence of causative pathogen from appropriately obtained specimens at the site of infection (eradication), repeat cultures were not performed/clinically indicated in a participant who had a clinical response of cure (presumed eradication) and detection of pathogen from the site of infection during therapy without need for antimicrobial treatment or a superinfection with a microbiological agent outside the treatment spectrum of ceftazidime-avibactam (gram positive/fungi) (colonization). 95% CI was based on Clopper-Pearson method.
Time Frame: Day 7 (from the data evaluated in approximately 21 months of the study)
Population: The microbiologically evaluable (ME) analysis set included all participants from the FAS with at least 72 hours use of ceftazidime-avibactam and at least 1 non-missing microbiological evaluation outcome. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 146
Percentage of Participants | 43.2 [35.0 to 51.6]

8. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Site Investigator at Day 14
Description: The microbiological success rate was defined as the number of participants with microbiological outcome "success" in a specific visit / number of participants with microbiological outcome assessed in a specific visit and was reported in terms of percentage of participants. Microbiological outcome as success was defined as absence of causative pathogen from appropriately obtained specimens at the site of infection (eradication), repeat cultures were not performed/clinically indicated in a participant who had a clinical response of cure (presumed eradication) and detection of pathogen from the site of infection during therapy without need for antimicrobial treatment or a superinfection with a microbiological agent outside the treatment spectrum of ceftazidime-avibactam (G+/fungi) (colonization). 95% CI was based on Clopper-Pearson method.
Time Frame: Day 14 (from the data evaluated in approximately 21 months of the study)
Population: The ME analysis set included all participants from the FAS with at least 72 hours use of ceftazidime-avibactam and at least 1 non-missing microbiological evaluation outcome. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 118
Percentage of Participants | 50.0 [40.7 to 59.3]

9. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Site Investigator at Day 21
Description: as for outcome 8
Time Frame: Day 21 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 85
Percentage of Participants | 49.4 [38.4 to 60.5]

10. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Site Investigator at Day 30
Description: as for outcome 8
Time Frame: Day 30 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 63
Percentage of Participants | 52.4 [39.4 to 65.1]

11. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Site Investigator at Day 60
Description: as for outcome 8
Time Frame: Day 60 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 28
Percentage of Participants | 64.3 [44.1 to 81.4]

12. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Site Investigator at EOT
Description: as for outcome 8
Time Frame: At EOT (maximum 86 days of treatment exposure) (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 202
Percentage of Participants | 69.8 [63.0 to 76.0]

13. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Central Laboratory at Day 7
Description: as for outcome 8
Time Frame: Day 7 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 165
Percentage of Participants | 46.1 [38.3 to 54.0]

14. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Central Laboratory at Day 14
Description: as for outcome 8
Time Frame: Day 14 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 126
Percentage of Participants | 50.0 [41.0 to 59.0]

15. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Central Laboratory at Day 21
Description: as for outcome 8
Time Frame: Day 21 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 90
Percentage of Participants | 54.4 [43.6 to 65.0]

16. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Central Laboratory at Day 30
Description: as for outcome 8
Time Frame: Day 30 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 69
Percentage of Participants | 49.3 [37.0 to 61.6]

17. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Central Laboratory at Day 60
Description: as for outcome 8
Time Frame: Day 60 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 29
Percentage of Participants | 65.5 [45.7 to 82.1]

18. Primary Outcome: Microbiological Success Rate Based on the Evaluation by Central Laboratory at EOT
Description: as for outcome 8
Time Frame: At EOT (maximum 86 days of treatment exposure) (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 207
Percentage of Participants | 69.6 [62.8 to 75.8]

19. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Site Investigator at Day 7
Description: as for outcome 8
Time Frame: Day 7 (from the data evaluated in approximately 21 months of the study)
Population: The ME analysis set included all participants from the FAS with at least 72 hours use of ceftazidime-avibactam and at least 1 non-missing microbiological evaluation outcome. All participants reported under, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure and contributed data to the table; however, may not have data evaluable for every row. ''Number Analyzed'' signifies participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 111
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 85
  Klebsiella pneumoniae | 43.5 [32.8 to 54.7]
  Pseudomonas aeruginosa: number analyzed (Participants) | 26
  Pseudomonas aeruginosa | 38.5 [20.2 to 59.4]

20. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Site Investigator at Day 14
Description: as for outcome 8
Time Frame: Day 14 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 90
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 71
  Klebsiella pneumoniae | 40.8 [29.3 to 53.2]
  Pseudomonas aeruginosa: number analyzed (Participants) | 19
  Pseudomonas aeruginosa | 42.1 [20.3 to 66.5]

21. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Site Investigator at Day 21
Description: as for outcome 8
Time Frame: Day 21 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 62
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 50
  Klebsiella pneumoniae | 46.0 [31.8 to 60.7]
  Pseudomonas aeruginosa: number analyzed (Participants) | 12
  Pseudomonas aeruginosa | 50.0 [21.1 to 78.9]

22. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Site Investigator at Day 30
Description: as for outcome 8
Time Frame: Day 30 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 43
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 35
  Klebsiella pneumoniae | 40.0 [23.9 to 57.9]
  Pseudomonas aeruginosa: number analyzed (Participants) | 8
  Pseudomonas aeruginosa | 50.0 [15.7 to 84.3]

23. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Site Investigator at Day 60
Description: as for outcome 8
Time Frame: Day 60 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 23
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 18
  Klebsiella pneumoniae | 66.7 [41.0 to 86.7]
  Pseudomonas aeruginosa: number analyzed (Participants) | 5
  Pseudomonas aeruginosa | 40.0 [5.3 to 85.3]

24. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Site Investigator at EOT
Description: as for outcome 8
Time Frame: At EOT (maximum 86 days of treatment exposure) (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 141
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 110
  Klebsiella pneumoniae | 65.5 [55.8 to 74.3]
  Pseudomonas aeruginosa: number analyzed (Participants) | 31
  Pseudomonas aeruginosa | 64.5 [45.4 to 80.8]

25. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Central Laboratory at Day 7
Description: as for outcome 8
Time Frame: Day 7 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 64
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 54
  Klebsiella pneumoniae | 44.4 [30.9 to 58.6]
  Pseudomonas aeruginosa: number analyzed (Participants) | 10
  Pseudomonas aeruginosa | 50.0 [18.7 to 81.3]

26. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Central Laboratory at Day 14
Description: as for outcome 8
Time Frame: Day 14 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 50
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 41
  Klebsiella pneumoniae | 29.3 [16.1 to 45.5]
  Pseudomonas aeruginosa: number analyzed (Participants) | 9
  Pseudomonas aeruginosa | 55.6 [21.2 to 86.3]

27. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Central Laboratory at Day 21
Description: as for outcome 8
Time Frame: Day 21 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 35
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 30
  Klebsiella pneumoniae | 46.7 [28.3 to 65.7]
  Pseudomonas aeruginosa: number analyzed (Participants) | 5
  Pseudomonas aeruginosa | 80.0 [28.4 to 99.5]

28. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Central Laboratory at Day 30
Description: as for outcome 8
Time Frame: Day 30 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 31
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 26
  Klebsiella pneumoniae | 30.8 [14.3 to 51.8]
  Pseudomonas aeruginosa: number analyzed (Participants) | 5
  Pseudomonas aeruginosa | 40.0 [5.3 to 85.3]

29. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Central Laboratory at Day 60
Description: as for outcome 8
Time Frame: Day 60 (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 15
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 13
  Klebsiella pneumoniae | 46.2 [19.2 to 74.9]
  Pseudomonas aeruginosa: number analyzed (Participants) | 2
  Pseudomonas aeruginosa | 100.0 [15.8 to 100.0]

30. Primary Outcome: Microbiological Success Rate by Pathogen Based on the Evaluation by Central Laboratory at EOT
Description: as for outcome 8
Time Frame: At EOT (maximum 86 days of treatment exposure) (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 74
Percentage of Participants
  Klebsiella pneumoniae: number analyzed (Participants) | 62
  Klebsiella pneumoniae | 64.5 [51.3 to 76.3]
  Pseudomonas aeruginosa: number analyzed (Participants) | 12
  Pseudomonas aeruginosa | 66.7 [34.9 to 90.1]

31. Primary Outcome: Number of Participants According to Indication for Ceftazidime-Avibactam at Index Date
Description: Index date was defined as the date when participants initiated >=1 dose of ceftazidime-avibactam treatment during the index hospitalization. Index hospitalization was defined as when participants' first hospitalization met the eligibility criteria.
Time Frame: At index date (from the data evaluated in approximately 21 months of the study)
Population: The FAS included all enrolled participants. The enrolled participants met the inclusion criteria, and did not meet the exclusion criteria. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 215
Participants
  Complicated intra-abdominal infections (cIAI) | 37
  Hospital-acquired pneumonia/ Ventilator-associated pneumonia (HAP/VAP) | 129
  Limited treatment options (LTO) | 49

32. Primary Outcome: Number of Participants According to Source of Infection
Description: as for outcome 31
Time Frame: At index date (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 174
Participants
  Hospital-acquired infection (HAI) | 134
  Community-acquired infection (CAI) | 40

33. Primary Outcome: Number of Isolated Strains
Description: The index date was defined as the date when participants initiated >=1 dose of ceftazidime-avibactam treatment during the index hospitalization. Index hospitalization was defined as when participants' first hospitalization met the eligible criteria.
Time Frame: At baseline (from 7 days prior to index date until index date) (from the data evaluated in approximately 21 months of the study)
Population: The FAS included all enrolled participants. The enrolled participants met the inclusion criteria, and did not meet the exclusion criteria. Here, ''Overall Number of Units Analyzed'' signifies number of strains evaluable for this outcome measure.
Measure: Number; unit: Strains
Units Other Than Participants: Strains
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Number analyzed (Strains) | 227
Strains
  Pseudomonas aeruginosa | 33
  Klebsiella pneumoniae | 129
  Serratia marcescens | 5
  Enterobacter cloacae | 4
  Escherichia coli | 4
  Proteus mirabilis | 3
  Klebsiella oxytoca | 1
  Other | 48

34. Primary Outcome: Number of Strains With Resistance to Ceftazidime-Avibactam and Other Antibiotic Drugs
Description: The index date was defined as the date when participants initiated >=1 dose of ceftazidime-avibactam treatment during the index hospitalization. Index hospitalization was defined as when participant's first hospitalization met the eligible criteria. Number of strains with resistance to ceftazidime-avibactam and other antibiotic drugs is reported. One strain could be resistant to more than one antibiotic.
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Number; unit: Strains
Units Other Than Participants: Strains
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 141
Number analyzed (Strains) | 162
Strains
  Klebsiella pneumoniae: Meropenem: number analyzed (Strains) | 116
  Klebsiella pneumoniae: Meropenem | 101
  Klebsiella pneumoniae: Imipenem: number analyzed (Strains) | 67
  Klebsiella pneumoniae: Imipenem | 58
  Klebsiella pneumoniae: Tigecycline: number analyzed (Strains) | 104
  Klebsiella pneumoniae: Tigecycline | 6
  Klebsiella pneumoniae: Ceftazidime-Avibactam: number analyzed (Strains) | 100
  Klebsiella pneumoniae: Ceftazidime-Avibactam | 5
  Klebsiella pneumoniae: Polymyxins: number analyzed (Strains) | 57
  Klebsiella pneumoniae: Polymyxins | 12
  Klebsiella pneumoniae: Polymyxin B: number analyzed (Strains) | 35
  Klebsiella pneumoniae: Polymyxin B | 3
  Pseudomonas aeruginosa: Meropenem: number analyzed (Strains) | 25
  Pseudomonas aeruginosa: Meropenem | 18
  Pseudomonas aeruginosa: Imipenem: number analyzed (Strains) | 16
  Pseudomonas aeruginosa: Imipenem | 13
  Pseudomonas aeruginosa: Tigecycline: number analyzed (Strains) | 14
  Pseudomonas aeruginosa: Tigecycline | 2
  Pseudomonas aeruginosa: Ceftazidime-Avibactam: number analyzed (Strains) | 22
  Pseudomonas aeruginosa: Ceftazidime-Avibactam | 1
  Pseudomonas aeruginosa: Polymyxins: number analyzed (Strains) | 12
  Pseudomonas aeruginosa: Polymyxins | 0
  Pseudomonas aeruginosa: Polymyxin B: number analyzed (Strains) | 7
  Pseudomonas aeruginosa: Polymyxin B | 0

35. Primary Outcome: Number of Carbapenem-Resistant Strains
Description: as for outcome 33
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Number; unit: Strains
Units Other Than Participants: Strains
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 134
Number analyzed (Strains) | 160
Strains
  Klebsiella pneumoniae | 108
  Pseudomonas aeruginosa | 25
  Enterobacter cloacae | 2
  Serratia marcescens | 3
  Escherichia coli | 4
  Other | 18

36. Secondary Outcome: Number of Participants According to Dose and Frequency of Ceftazidime-Avibactam: Full Analysis Set
Description: Frequency of Ceftazidime-Avibactam was divided into: BID = Bis in die (twice a day), TID = Ter in die (thrice a day) and QD = Quaque die (once a day). A participant who had more than one record of treatment within the same dosage and frequency was counted only once.
Time Frame: From start of index treatment to end of index treatment (maximum 86 days of treatment exposure) (from the data evaluated in approximately 21 months of the study)
Population: The FAS included all enrolled participants. The enrolled participants met the inclusion criteria, and did not meet the exclusion criteria. Here, ''Number Analyzed'' signifies participants evaluable for the specified dosage. All participants under "Number of Participants Analyzed" contributed data to the table but may not have evaluable data for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Participants
  2.5 grams: TID: number analyzed (Participants) | 206
  2.5 grams: TID | 178
  2.5 grams: BID: number analyzed (Participants) | 206
  2.5 grams: BID | 18
  2.5 grams: QD: number analyzed (Participants) | 206
  2.5 grams: QD | 8
  2.5 grams: Other: number analyzed (Participants) | 206
  2.5 grams: Other | 10
  1.25 grams: TID: number analyzed (Participants) | 21
  1.25 grams: TID | 15
  1.25 grams: BID: number analyzed (Participants) | 21
  1.25 grams: BID | 7
  1.25 grams: QD: number analyzed (Participants) | 21
  1.25 grams: QD | 1
  1.25 grams: Other: number analyzed (Participants) | 21
  1.25 grams: Other | 2
  0.94 grams: QD: number analyzed (Participants) | 1
  0.94 grams: QD | 1
  1 gram: BID: number analyzed (Participants) | 1
  1 gram: BID | 1
  2 grams: TID: number analyzed (Participants) | 1
  2 grams: TID | 1
  3 grams: BID: number analyzed (Participants) | 1
  3 grams: BID | 1

37. Secondary Outcome: Number of Participants According to Dose and Frequency of Ceftazidime-Avibactam: Clinically Evaluable Analysis Set
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Participants
  2.5 grams: TID: number analyzed (Participants) | 200
  2.5 grams: TID | 173
  2.5 grams: BID: number analyzed (Participants) | 200
  2.5 grams: BID | 17
  2.5 grams: QD: number analyzed (Participants) | 200
  2.5 grams: QD | 8
  2.5 grams: Other: number analyzed (Participants) | 200
  2.5 grams: Other | 10
  1.25 grams: TID: number analyzed (Participants) | 21
  1.25 grams: TID | 15
  1.25 grams: BID: number analyzed (Participants) | 21
  1.25 grams: BID | 7
  1.25 grams: QD: number analyzed (Participants) | 21
  1.25 grams: QD | 1
  1.25 grams: Other: number analyzed (Participants) | 21
  1.25 grams: Other | 2
  0.94 grams: QD: number analyzed (Participants) | 1
  0.94 grams: QD | 1
  1 gram: BID: number analyzed (Participants) | 1
  1 gram: BID | 1
  2 grams: TID: number analyzed (Participants) | 1
  2 grams: TID | 1
  3 grams: BID: number analyzed (Participants) | 1
  3 grams: BID | 1

38. Secondary Outcome: Duration of Exposure to Ceftazidime-Avibactam: Full Analysis Set
Description: For a participant, each ceftazidime-avibactam administration period (days) was calculated as: ceftazidime-avibactam administration end date - ceftazidime-avibactam administration start date + 1. Duration of exposure (days) was obtained by summing up all ceftazidime-avibactam administration periods.
Time Frame: as for outcome 36
Population: The FAS included all enrolled participants. The enrolled participants met the inclusion criteria, and did not meet the exclusion criteria.
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Days | 12.0 [2 to 86]

39. Secondary Outcome: Duration of Exposure to Ceftazidime-Avibactam: Clinically Evaluable Analysis Set
Description: as for outcome 38
Time Frame: as for outcome 36
Population: as for outcome 6
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Days | 12.0 [3 to 86]

40. Secondary Outcome: Number of Participants Who Received Combination Therapy With Ceftazidime-Avibactam: Full Analysis Set
Time Frame: as for outcome 36
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Participants | 176

41. Secondary Outcome: Number of Participants Who Received Combination Therapy With Ceftazidime-Avibactam: Clinically Evaluable Analysis Set
Time Frame: as for outcome 36
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Participants | 172

42. Secondary Outcome: Hospital Length of Stay (LOS): Full Analysis Set
Description: Hospital LOS was defined as date of hospital discharge minus date of hospital admission plus 1. The index date was defined as the date when participants initiated >=1 dose of ceftazidime-avibactam treatment during the index hospitalization. Index hospitalization was defined as when participants' first hospitalization met the eligible criteria.
Time Frame: From index date up to hospital discharge, in-hospital death, withdrawal from study, or lost to follow-up, whichever occurred first (approximately 27 months including 6 months of index period); (from data evaluated in approximately 21 months of the study)
Population: as for outcome 38
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Days | 36.5 [4 to 751]

43. Secondary Outcome: Hospital Length of Stay (LOS): CE Analysis Set
Description: as for outcome 42
Time Frame: as for outcome 42
Population: as for outcome 6
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Days | 36.0 [6 to 751]

44. Secondary Outcome: Intensive Care Unit (ICU) LOS: Full Analysis Set
Description: Duration of ICU stay was defined as date of ICU discharge minus date of ICU admission plus 1. The index date was defined as the date when participants initiated >=1 dose of ceftazidime-avibactam treatment during the index hospitalization. Index hospitalization was defined as when participants' first hospitalization met the eligible criteria.
Time Frame: During index hospitalization, approximately 27 months including 6 months of index period; (from the data evaluated in approximately 21 months of the study)
Population: The FAS included all enrolled participants. The enrolled participants met the inclusion criteria, and did not meet the exclusion criteria. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 99
Days | 25.0 [1 to 751]

45. Secondary Outcome: ICU LOS: Clinically Evaluable Analysis Set
Description: as for outcome 44
Time Frame: as for outcome 44
Population: The CE analysis set included all participants from the FAS with at least 72 hours use of ceftazidime-avibactam and at least 1 non-missing clinical evaluation outcome. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 95
Days | 25.0 [1 to 751]

46. Secondary Outcome: Number of Participants According to Most Frequent Diagnosis at Admission: Full Analysis Set
Description: The number of participants reported according to the most frequent diagnosis at admission to the hospital were reported in this outcome measure.
Time Frame: At admission to the hospital (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Participants
  Pneumonia | 31
  Respiratory failure | 29
  Hypertension | 24

47. Secondary Outcome: Number of Participants According to Most Frequent Diagnosis at Admission: Clinically Evaluable Analysis Set
Description: as for outcome 46
Time Frame: At admission to the hospital (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Participants
  Pneumonia | 31
  Respiratory failure | 29
  Hypertension | 23

48. Secondary Outcome: Number of Participants According to Most Frequent Diagnosis at Discharge: Full Analysis Set
Description: The number of participants reported according to the most frequent diagnosis at discharge from the hospital were reported in this outcome measure.
Time Frame: At discharge from the hospital (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Participants
  Pneumonia | 121
  Septic shock | 42
  Sepsis | 39

49. Secondary Outcome: Number of Participants According to Most Frequent Diagnosis at Discharge: Clinically Evaluable Analysis Set
Description: as for outcome 48
Time Frame: At discharge from the hospital (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Participants
  Pneumonia | 120
  Septic shock | 42
  Sepsis | 39

50. Secondary Outcome: Number of Participants With at Least 1 Concomitant Procedures: Full Analysis Set
Description: The number of participants with at least 1 concomitant procedure were reported in this outcome measure. The index date was defined as the date when participants initiated >=1 dose of ceftazidime-avibactam treatment during the index hospitalization. Index hospitalization was defined as when participants' first hospitalization met the eligible criteria.
Time Frame: From start of index treatment until death, withdraw of the study, 60 days following hospital discharge, whichever comes first (approximately 27 months including 6 months of index period); (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Participants | 193

51. Secondary Outcome: Number of Participants With at Least 1 Concomitant Procedures: Clinically Evaluable Analysis Set
Description: as for outcome 50
Time Frame: as for outcome 50
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Participants | 187

52. Secondary Outcome: Duration of Mechanical Ventilation: Full Analysis Set
Description: For a participant, each mechanical ventilation period (days) was calculated as: mechanical ventilation end date - mechanical ventilation start date + 1. Length of mechanical ventilation (days) was obtained by summing up all mechanical ventilation periods. The index date was defined as the date when participants initiated >=1 dose of ceftazidime-avibactam treatment during the index hospitalization. Index hospitalization was defined as when participants' first hospitalization met the eligible criteria.
Time Frame: as for outcome 50
Population: as for outcome 31
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 72
Days | 17.0 [1 to 128]

53. Secondary Outcome: Duration of Mechanical Ventilation: Clinically Evaluable Analysis Set
Description: as for outcome 52
Time Frame: as for outcome 50
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 71
Days | 17.0 [1 to 128]

54. Secondary Outcome: Percentage of Participants With Readmission Due to Recurrence of Infection Within 30 Days and 31-60 Days After Discharge: Full Analysis Set
Description: 95% CI was based on Clopper-Pearson method.
Time Frame: Within 30 days and 31-60 days after discharge (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Percentage of Participants
  Within 30 days after discharge | 10 [6 to 15]
  Within 31-60 days after discharge | 3 [1 to 6]

55. Secondary Outcome: Percentage of Participants With Readmission Due to Recurrence of Infection Within 30 Days and 31-60 Days After Discharge: CE Analysis Set
Description: 95% CI was based on Clopper-Pearson method.
Time Frame: Within 30 days and 31-60 days after discharge (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Percentage of Participants
  Within 30 days after discharge | 10 [7 to 15]
  Within 31-60 days after discharge | 3 [1 to 6]

56. Secondary Outcome: Percentage of Participants Who Died During Hospitalization: Full Analysis Set
Description: In hospital-mortality was defined as deaths occurring after treatment initiation but before hospital discharge. The percentage of participants who died during index hospitalization were reported in this outcome measure. Index hospitalization was defined as when participants' first hospitalization met the eligible criteria. 95% CI was based on Clopper-Pearson method.
Time Frame: During index hospitalization (approximately 27 months including 6 months of index period); (from the data evaluated in approximately 21 months of the study)
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 220
Percentage of Participants | 10 [6 to 15]

57. Secondary Outcome: Percentage of Participants Who Died During Hospitalization: Clinically Evaluable Analysis Set
Description: as for outcome 56
Time Frame: as for outcome 56
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftazidime-Avibactam
Number analyzed (Participants) | 214
Percentage of Participants | 10 [6 to 15]

ADVERSE EVENTS:
Time Frame: From index date up to 60 days after hospital discharge, in-hospital death, withdrawal from the study, or lost to follow-up, whichever occurred first (approximately 27 months including 6 months of index period); (from the data evaluated in approximately 21 months of the study)
Description: The index date was defined as the date when participants initiated >=1 dose of ceftazidime-avibactam treatment during the index hospitalization. Index hospitalization was defined as when participants' first hospitalization met the eligible criteria. The FAS included all enrolled participants. The enrolled participants met the inclusion criteria, and did not meet the exclusion criteria.
Arm/Group | Ceftazidime-Avibactam
All-Cause Mortality (participants affected / at risk) | 22/220
Serious Adverse Events (participants affected / at risk) | 0/220
Other Adverse Events (participants affected / at risk) | 0/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT05487586/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT05487586/SAP_001.pdf